CLINICAL TRIAL: NCT06063785
Title: Multispectral Optoacoustic Tomography for the Assessment of Liver Fibrosis and Gastrointestinal Transit in Patients With Cystic Fibrosis
Brief Title: Multispectral Optoacoustic Tomography in Patients With Cystic Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Adrian Regensburger (Unknown)
Responsible Party: Principal Investigator, Alexander Schnell, Principal Investigator, University of Erlangen-Nürnberg Medical School
Other Study IDs: CF_MSOT
Record Dates: First submitted 2023-09-05; First posted 2023-10-03 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Cystic Fibrosis; Liver Fibrosis; Gastrointestinal Transport Disorder; Dios
Keywords: Cystic Fibrosis; MSOT; Liver Fibrosis; Gastrointestinal Transit
MeSH Terms: conditions — Cystic Fibrosis; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples for bile acid profiling Stool samples for bile acid profiling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CF with liver affection: CF patients with proven CF hepatopathy
  Interventions: Diagnostic Test: Acoustic Radiation Forced Impulse Imaging; Diagnostic Test: Multispectral Optoacoustic Tomography
- CF without liver affection: CF patients without proven CF hepatopathy
  Interventions: Diagnostic Test: Acoustic Radiation Forced Impulse Imaging; Diagnostic Test: Multispectral Optoacoustic Tomography
- Healthy volunteers: Healthy volunteers without liver affection
  Interventions: Diagnostic Test: Acoustic Radiation Forced Impulse Imaging; Diagnostic Test: Multispectral Optoacoustic Tomography

INTERVENTIONS:
Diagnostic Test: Acoustic Radiation Forced Impulse Imaging — Measurement of Liver stiffness
  Other Names: ARFI
Diagnostic Test: Multispectral Optoacoustic Tomography — Measurement of optoacoustic spectra in liver and gastrointestinal tract
  Other Names: MSOT

SUMMARY:
Cystic fibrosis (CF) is the most common hereditary disease in Central Europe. The disease is caused by a mutation in the cystic fibrosis transmembrane conductance regulator gene (CFTR). In the liver, fibrotic remodeling can lead to liver cirrhosis in the long term. Early detection of CF hepatopathy is essential to therapeutically slow down the progression of fibrotic remodeling mechanisms. Newborns suffering from CF have a significantly increased risk for the occurrence of meconium ileus and also with advancing age there are symptoms ranging from chronic constipation to Distal Intestinal Obstruction Syndrome (DIOS), due to a reduction of intestinal motility.

In this study, the degree of liver fibrosis will now be investigated in adult patients with cystic fibrosis using Multispectral Optoacoustic Imaging (MSOT). In addition, gastrointestinal passage will be studied non-invasively to investigate another affection of the gastrointestinal system.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is the most common hereditary disease in Central Europe, with an incidence of approximately 3,300 to 4,800 new cases. The disease follows an autosomal recessive pattern of inheritance, the cause being a mutation in the cystic fibrosis transmembrane conductance regulator gene (CFTR). In the liver, fibrotic remodeling can lead to liver cirrhosis in the long term. Early detection of CF hepatopathy is essential to therapeutically slow down the progression of fibrotic remodeling mechanisms. Over the past decade, measurements of liver stiffness using Acoustic Radiation Force Impulse Imaging (ARFI) have proven to be a valid tool for measuring fibrotic tissue remodeling in CF in adults and children. Furthermore, in the gastrointestinal tract, serious consequences result from the absence of the CFTR channel. Newborns suffering from CF have a significantly increased risk for the occurrence of meconium ileus and also with advancing age there are symptoms ranging from chronic constipation to DIOS (Distal Intestinal Obstruction Syndrome), due to a reduction of intestinal motility.

By means of new imaging methods, such as multispectral optoacoustic tomography, it is possible to examine not only the body's own substances but also substances foreign to the body. With Multispectral Optoacoustic Imaging (MSOT), similar to conventional sonography, a transducer is placed on the skin and instead of sound, energy is applied to the tissue by means of light flashes. This leads to a constant alternation of minimal expansions and contractions (thermoelastic expansion) of individual tissue components or molecules. Previous studies have shown that quantitative determination of hemoglobin can provide information on blood flow and inflammatory activity in the intestines of adult patients with Crohn's disease. Also, fibrotic changes in the liver can probably be detected with this method, similar to that in muscle tissue. Furthermore, we have recently shown that orally ingested Indocyanine green (ICG) can be detected in the small intestine and thus conclusions can be drawn about gastrointestinal passage, without the use of ionizing radiation. In this study, the degree of liver fibrosis will now be investigated in adult patients with cystic fibrosis using MSOT. In addition, gastrointestinal passage will be studied non-invasively to investigate another affection of the gastrointestinal system.

ELIGIBILITY:
Inclusion Criteria:

Patient cohort "Cystic Fibrosis without CF-related liver disease":

* Molecular genetic confirmed diagnosis of cystic fibrosis.
* Age over 18 years
* Written informed consent

Patient cohort "Cystic Fibrosis with CF-related liver disease":

* Molecular genetic confirmed diagnosis of cystic fibrosis
* Presence of CF-related liver disease based on Colombo criteria:

  * Hepato- and/or splenomegaly
  * Persistent elevation of transaminases in the serum
  * Sonographic evidence of liver involvement
* Age over 18 years
* Written informed consent

"Volunteer Subjects":

* Age over 18 years
* Written informed consent

Exclusion Criteria:

General:

* Pregnancy
* Breastfeeding mothers
* Tattoo in the area of the examination
* Subcutaneous fat tissue over 3 cm

Patient cohort "Cystic fibrosis without CF-related liver disease":

* Taking systemic glucocorticoids or immunosuppressants as part of a permanent medication regimen.
* Presence of CF-related liver disease based on Colombo criteria:

  * Hepato- and/or splenomegaly.
  * Persistent elevation of transaminases in the serum
  * Sonographic evidence of liver involvement.
* Acute exacerbation of infection

Patient cohort "Cystic fibrosis with CF-related liver disease":

* Taking systemic glucocorticoids or immunosuppressants as part of a permanent medication regimen.
* Decompensation of CF-related liver disease
* Acute exacerbation of infection

"volunteer subjects":

* Presence of liver disease
* Use of systemic glucocorticoids or immunosuppressants in the context of permanent medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is planned to study a total of 10 patients each with cystic fibrosis with/without CF-related liver disease and 10 healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Quantitative collagen signal (Liver) | Day 1
  in arbitrary units
Quantitative Indocyanine Green (ICG) signal (Intestinal) | 0, 60, 90, 120, 180, 240, 300min post ICG intake
  Day 1

SECONDARY OUTCOMES:
Quantitative oxy/deoxygenated hemoglobin signal (Liver) | Day 1
  in arbitrary units
Quantitative oxy/deoxygenated hemoglobin signal (Intestinal) | 0, 60, 90, 120, 180, 240, 300min post ICG intake
  in arbitrary units
Quantitative single wave lengths (Intestinal) | 0, 60, 90, 120, 180, 240, 300min post ICG intake
  in arbitrary units
Quantitative single wave lengths (Liver) | Day 1
  in arbitrary units
Optoacoustic spectrum (Intestinal) | 0, 60, 90, 120, 180, 240, 300min post ICG intake
  in arbitrary units, normalized
Optoacoustic spectrum (Liver) | Day 1
  in arbitrary units, normalized
Shear wave velocity (Liver) | Day 1
  in m/s
Attenuation coefficient (Liver) | Day 1
  in dB/cm/MHz
Chenodeoxycholic acid (CDCA) and respective glycine and taurine conjugates | Day 1
  µmol/l and /g stool
Cholic acid (CA) and respective glycine and taurine conjugates | Day 1
  µmol/l and /g stool
Deoxycholic acid (DCA) and respective glycine and taurine conjugates | Day 1
  µmol/l and /g stool
Lithocholic acid (LCA) and respective glycine and taurine conjugates | Day 1
  µmol/l and /g stool
Ursodeoxycholic acid (UDCA) and respective glycine and taurine conjugates | Day 1
  µmol/l and /g stool

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Schnell, Principal Investigator — Department of Pediatric and Adolescent Medicine, University Hospital Erlangen; Adrian P Regensburger, Principal Investigator — Department of Pediatric and Adolescent Medicine, University Hospital Erlangen
Locations (1):
- University Hospital Erlange, Department of Pediatrics, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No